CLINICAL TRIAL: NCT01210690
Title: Observational Sentinel Sites Study in Infants Younger Than 12 Months Who Are Prescribed Treatment With Keppra® (Levetiracetam) Oral Solution in Usual Clinical Practice
Brief Title: Observational Study in Infants Who Are Prescribed Treatment With Keppra® (Levetiracetam) Oral Solution
Status: Completed | Type: Observational
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: N01357; 2009-017333-21 (EudraCT Number)
Record Dates: First submitted 2010-09-23; First posted 2010-09-28 (Estimated); Results first posted 2014-11-19 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Epilepsy
Keywords: Levetiracetam; Keppra® Oral Solution; Keppra® in Children
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients, 1 - 11 months old, prescribed Keppra® oral solution: Epileptic patients who have been prescribed Keppra® (Levetiracetam) oral solution and who are between 1 and 11 months old. The patients will be followed as per current clinical practices for their condition. The choice of medical treatment, including the concomitant use of other antiepileptic drugs, is made independently by the physician in the regular course of practice and is not influenced by the study protocol.

SUMMARY:
The purpose of this observational study is to broaden the knowledge of the known safety and efficacy profile of Keppra® (Levetiracetam) oral solution in epileptic infants younger than 12 months when treated according to routine clinical practice. Their data will be collected until they reach the age of 13 months.

DETAILED DESCRIPTION:
This non-interventional sentinel sites post-authorization safety study (PASS) aims to collect additional data on use of Keppra® (Levetiracetam) oral solution in clinical practice, and on efficacy and safety of Keppra® (Levetiracetam) in infants younger than12 months. Epileptic patients between the age of 1 month and 11 months inclusive can be invited for participation to the non-interventional sentinel sites PASS, after the physician has decided to initiate therapy with Keppra® (Levetiracetam) oral solution (100 mg/ml bottle) and patient has so far been treated with Keppra® (Levetiracetam) for no longer than 10 days. The patients will be followed and their data will be collected until they reach the age of 13 months.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of epilepsy
* being treated with Keppra® Oral Solution
* aged between 1 month and 11 months inclusive at study baseline

Exclusion Criteria:

* none

Ages: 1 Month to 11 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients coming to day clinic for consultation by specialist
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2011-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (27):
- France (3):
  - 012, Amiens
  - 010, Bron
  - 011, Paris
- Germany (6):
  - 027, Berlin
  - 024, Bielefeld
  - 026, Heidelberg
  - 021, Kehl Kork
  - 023, Kiel
  - 022, Münster
- Greece (2):
  - 072, Athens
  - 071, Pátrai
- Italy (5):
  - 037, Bologna
  - 031, Calambrone
  - 032, Milan
  - 034, Roma
  - 035, Verona
- Poland (4):
  - 065, Gdansk
  - 064, Lodz
  - 063, Szczecin
  - 062, Warsaw
- Spain (4):
  - 043, Barcelona
  - 044, Madrid
  - 045, Madrid
  - 046, Murcia
- United Kingdom (3):
  - 057, Birmingham
  - 052, Liverpool
  - 051, London

REFERENCES:
- See also: FDA safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: It was planned to enroll 100 patients at approximately 30-40 sites in the European Union.
Pre-assignment Details: Overall 101 patients were enrolled. The Participant Flow refers to the Enrolled Set (ES). The ES consisted of patients with a signed Data Consent Form.
Groups:
- Patients, 1 - 11 Months Old, Prescribed Keppra® Oral Solution: Epileptic patients who have been prescribed Keppra® (Levetiracetam) oral solution and who were between 1 and 11 months old. The patients were followed as per current clinical practices for their condition. The choice of medical treatment, including the concomitant use of other antiepileptic drugs, was made independently by the physician in the regular course of practice and was not influenced by the study protocol.
Period: Overall Study
Arm/Group | Patients, 1 - 11 Months Old, Prescribed Keppra® Oral Solution
Started | 101
Completed | 75
Not Completed | 26
Not completed — Adverse Event | 7
Not completed — Lack of Efficacy | 12
Not completed — Lost to Follow-up | 3
Not completed — Disease Remission | 1
Not completed — Withdrawal by Subject | 1
Not completed — Patient refused to swallow | 1
Not completed — Patient could not take glucose | 1

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population refers to the Safety Set (SS). The SS consisted of all patients in the Enrolled Set who received at least 1 (partial) dose of study medication.
Arm/Group | Patients, 1 - 11 Months Old, Prescribed Keppra® Oral Solution
Number analyzed (Participants) | 101
Age, Continuous [Mean (Standard Deviation); unit: months] | 6.0 (3.0)
Age, Customized [Number; unit: participants]
  <1 month | 2
  ≥1 - ≤6 months | 53
  ≥6 - ≤11 months | 46
  >11 months | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 50
Weight [Mean (Standard Deviation); unit: kilogram] | 7.00 (1.94)
Height [Mean (Standard Deviation); unit: centimeter] | 64.16 (8.04)

OUTCOME MEASURES:

1. Primary Outcome: Treatment-Emergent Adverse Events (TEAEs) From Baseline Through Safety Follow-up Visit
Description: Number of patients with any Treatment-Emergent Adverse Events (TEAEs) as reported by the patient's parent and/or caregiver or observed by the treating physician during the study (maximum Treatment Period is 12 months plus 2-week safety follow-up).
Time Frame: From Baseline through the Safety Follow-up Visit (maximum Treatment Period is 12 months plus 2-week safety follow-up)
Population: The Analysis Population refers to the Safety Set (SS). The SS consisted of all patients in the Enrolled Set who received at least 1 (partial) dose of study medication.
Measure: Number; unit: participants
Arm/Group | Patients, 1 - 11 Months Old, Prescribed Keppra® Oral Solution
Number analyzed (Participants) | 101
participants | 55

2. Secondary Outcome: Incidence of Overall Serious Treatment-Emergent Adverse Events (TEAEs) From Baseline Through the Safety Follow-up
Description: Number of patients with any serious Treatment-Emergent Adverse Events (TEAEs) during the study (maximum Treatment Period is 12 months plus 2-week safety follow-up).
Time Frame: From Baseline through the Safety Follow-up Visit (maximum Treatment Period is 12 months plus 2-weeks safety follow-up)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Patients, 1 - 11 Months Old, Prescribed Keppra® Oral Solution
Number analyzed (Participants) | 101
participants | 32

3. Secondary Outcome: Incidence of Treatment-Emergent Adverse Events (TEAEs) Leading to Temporary or Permanent Discontinuation of Keppra® (Levetiracetam) From Baseline Through the Last Visit
Description: Number of patients with any Treatment-Emergent Adverse Events (TEAEs) leading to temporary or permanent discontinuation of Keppra® (Levetiracetam) during the Treatment Period (maximum 12 months).
Time Frame: From Baseline through the last Treatment Visit (maximum 12 months)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Patients, 1 - 11 Months Old, Prescribed Keppra® Oral Solution
Number analyzed (Participants) | 101
participants | 5

4. Secondary Outcome: Presence of Deviation From the Normal Milestones of Psychomotor Development From Baseline to the Last Treatment Visit
Description: Number of patients with presence of deviation from the normal milestones of psychomotor development during the Treatment Period (maximum 12 months). The treating physician evaluated at each visit, as part of standard clinical practice, the psychomotor development of the patient. The evaluation of the patient's psychomotor development was categorized by the motor development, the social development and the language development.
Time Frame: From Baseline to the last Treatment Visit (maximum 12 months)
Population: The Analysis Population refers to the Safety Set (SS). The SS consisted of all patients in the Enrolled Set who received at least 1 (partial) dose of study medication. Presented is the number of subjects with non-missing data on psychomotor development at the corresponding visit.
Measure: Number; unit: participants
Arm/Group | Patients, 1 - 11 Months Old, Prescribed Keppra® Oral Solution
Number analyzed (Participants) | 81
participants
  Any deviation | 54
  Motor development | 52
  Social development | 48
  Language development | 48

5. Secondary Outcome: Mean Change From Baseline in Standardized Body Weight Scores at the Safety Follow-up Visit
Description: For each visit, body weight was measured and standardization for gender and age was performed based on WHO growth charts to obtain z-scores. For this outcome measure, the mean of the differences of individual body weight z-scores from Safety Follow-up Visit to Baseline was determined.
Time Frame: From Baseline to the safety follow-up visit (maximum treatment period is 12 months plus 2-week safety follow-up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: z-scores
Arm/Group | Patients, 1 - 11 Months Old, Prescribed Keppra® Oral Solution
Number analyzed (Participants) | 18
z-scores | 0.740 (1.304)

6. Secondary Outcome: Mean Change From Baseline in Standardized Body Length Scores at the Safety Follow-up Visit
Description: For each visit, body length was measured and age standardization was performed based on WHO growth charts to obtain z-scores. For this outcome measure, the difference of body length z-scores from Safety Follow-up Visit to Baseline was determined and averaged across the study population.
Time Frame: From Baseline to the Safety Follow-up Visit (maximum Treatment Period is 12 months plus 2-week safety follow-up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: z-scores
Arm/Group | Patients, 1 - 11 Months Old, Prescribed Keppra® Oral Solution
Number analyzed (Participants) | 15
z-scores | 0.335 (2.058)

7. Secondary Outcome: Mean Change From Baseline in Standardized Head Circumference Scores at the Safety Follow-up Visit
Description: For each visit, head circumference was measured and age standardization was performed based on WHO growth charts to obtain z-scores. For this outcome measure, the difference of head circumference z-scores from Safety Follow-up Visit to Baseline was determined and averaged across the study population.
Time Frame: From Baseline to the Safety Follow-up Visit (maximum Treatment Period is 12 months plus 2-week safety follow-up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: z-scores
Arm/Group | Patients, 1 - 11 Months Old, Prescribed Keppra® Oral Solution
Number analyzed (Participants) | 15
z-scores | -0.307 (1.802)

8. Secondary Outcome: Number of Patients With Abnormalities Noted During Physical Examination From Baseline to the Last Treatment Visit
Description: Number of patients with abnormalities noted during physical examination over the Treatment Period (maximum 12 months). Any abnormal findings during the physical examination during the study were reported as Adverse Events (AEs).
  The Number of Patients With Abnormalities Noted During Physical Examination From Baseline to the Last Treatment Visit cannot be given because abnormalities at Screening are listed only and worsening after Screening were handled as AEs and tabulated along with the other AEs.
Time Frame: From Baseline to the last Treatment Visit (maximum 12 months)
Reporting Status: Not Posted

9. Secondary Outcome: Number of Patients With Abnormalities Noted During Neurological Examination From Baseline to the Last Treatment Visit
Description: The Number of Patients With Abnormalities Noted During Neurological Examination cannot be given because abnormality frequencies were only determined for single parameters of the neurological examination and therefore a subject might have been counted several times.
Time Frame: From Baseline to the last Treatment Visit (maximum 12 months)
Reporting Status: Not Posted

10. Secondary Outcome: Global Evaluation Scale of the Psychomotor Development (GES)
Description: Global evaluation scale of the psychomotor development (GES): physician's assessment of the change from Baseline in the psychomotor development at the last Treatment Visit (maximum timeframe is 12 months). The GES is a 7-point scale with the following options:
  7=Marked improvement
  6=Moderate improvement
  5=Slight improvement
  4=No Change
  3=Slight worsening
  2=Moderate worsening
  1=Marked worsening
  As a variant of this variable, a 3-class variable was derived as follows
  * "Marked improvement," "Moderate improvement," and "Slight improvement" were defined as "Improved."
  * "No change" was defined as "Stable."
  * "Slight worsening," "Moderate worsening," and "Marked worsening" were defined as "Worsened."
Time Frame: From Baseline to the last Treatment Visit (maximum 12 months)
Population: The Analysis Population refers to the Full Analysis Set (FAS). The FAS consisted of all patients in the Enrolled Set who had at least 1 post-Baseline efficacy assessment. Presented is the number of subjects with a non-missing measurement at Visit 7.
Measure: Number; unit: participants
Arm/Group | Patients, 1 - 11 Months Old, Prescribed Keppra® Oral Solution
Number analyzed (Participants) | 85
participants
  Improved | 45
  Stable | 31
  Worsened | 9

11. Secondary Outcome: Global Evaluation Scale of Epilepsy Severity (GES)
Description: Global evaluation scale of epilepsy severity (GES): physician's assessment of the change from Baseline of the epilepsy severity at the last Treatment Visit (maximum 12 months). The GES is a 7-point scale that assesses change in the severity of the patient's illness. The GES is a 7-point scale with the following options:
  7=Marked improvement
  6=Moderate improvement
  5=Slight improvement
  4=No Change
  3=Slight worsening
  2=Moderate worsening
  1=Marked worsening
  As a variant of this variable, a 3-class variable was derived as follows
  * "Marked improvement," "Moderate improvement," and "Slight improvement" were defined as "Improved."
  * "No change" was defined as "Stable."
  * "Slight worsening," "Moderate worsening," and "Marked worsening" were defined as "Worsened."
Time Frame: From Baseline to the last Treatment Visit (maximum time frame is 12 months)
Population: as for outcome 10
Measure: Number; unit: participants
Groups:
- Patients, 1 - 11 Months Old, Prescribed Keppra® Oral Solution: Epileptic patients who have been prescribed Keppra® (Levetiracetam) oral solution and who were between 1 and 11 months old. The patients were followed as per current clinical practices for their condition. The choice of medical treatment, including the concomitant use of other antiepileptic drugs, was made independently by the physician in the regular course of practice and is not influenced by the study protocol.
Arm/Group | Patients, 1 - 11 Months Old, Prescribed Keppra® Oral Solution
Number analyzed (Participants) | 85
participants
  Improved | 61
  Stable | 16
  Worsened | 8

12. Secondary Outcome: Number of Patients Who Withdraw Due to Lack or Loss of Efficacy During the Treatment Period
Description: Number of patients who withdraw due to lack or loss of efficacy during the Treatment Period (maximum 12 months).
Time Frame: From Baseline through the last Treatment Visit (maximum 12 months)
Population: The Analysis Population refers to the Full Analysis Set (FAS). The FAS consisted of all patients in the Enrolled Set who had at least 1 post-Baseline efficacy assessment.
Measure: Number; unit: participants
Arm/Group | Patients, 1 - 11 Months Old, Prescribed Keppra® Oral Solution
Number analyzed (Participants) | 101
participants | 12

ADVERSE EVENTS:
Time Frame: Treatment emergent Adverse Events (TEAEs) were reported from Baseline through the Safety Follow-up Visit.
Description: Treatment emergent Adverse Events (AEs) are AEs with onset date (including severity-worsening) on or after first dose of study medication.
Groups:
- Patients, 1 - 11 Mths Old, Prescribed Keppra® Oral Solution: Epileptic patients who have been prescribed Keppra® (Levetiracetam) oral solution and who were between 1 and 11 months old. The patients were followed as per current clinical practices for their condition. The choice of medical treatment, including the concomitant use of other antiepileptic drugs, was made independently by the physician in the regular course of practice and was not influenced by the study protocol.
Arm/Group | Patients, 1 - 11 Mths Old, Prescribed Keppra® Oral Solution
Serious Adverse Events (participants affected / at risk) | 32/101
Other Adverse Events (participants affected / at risk) | 19/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients, 1 - 11 Mths Old, Prescribed Keppra® Oral Solution (N=101)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (3)
Drug withdrawal syndrome (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Bronchiolitis (Infections and infestations) | 2 (2)
Bronchitis (Infections and infestations) | 2 (2)
Gastroenteritis (Infections and infestations) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 2 (3)
Candida infection (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Convulsion (Nervous system disorders) | 10 (15)
Epilepsy (Nervous system disorders) | 3 (5)
Hydrocephalus (Nervous system disorders) | 1 (1)
Hyperkinesia (Nervous system disorders) | 1 (1)
Infantile spasms (Nervous system disorders) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (1)
Inappropriate affect (Psychiatric disorders) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Neurosurgery (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients, 1 - 11 Mths Old, Prescribed Keppra® Oral Solution (N=101)
Diarrhoea (Gastrointestinal disorders) | 6 (8)
Pyrexia (General disorders) | 7 (8)
Bronchitis (Infections and infestations) | 9 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days